CLINICAL TRIAL: NCT02971150
Title: Treatment Resistant Depression and Insomnia in Older Veterans: A Pilot Study
Brief Title: Treatment Resistant Depression and Insomnia in Older Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PRO0001567
Record Dates: First submitted 2016-11-17; First posted 2016-11-22 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Treatment Resistant Depression; Insomnia
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BBTI (Experimental): Participants will receive Brief Behavioral Treatment for Insomnia (BBTI). This will be administered over the course of 4 weeks. BBTI is based on the concepts of sleep restriction and stimulus control. The first and third session are in person and the 2 and 4th session are conducted over the phone. Throughout the treatment, participants will complete daily sleep dairies. After 4 weeks of treatment, participants randomized to this group will cross over to the no intervention group and will be called once a week to assess mood and sleep symptoms.
  Interventions: Behavioral: Brief Behavioral Treatment for Insomnia
- Control (No Intervention): Participants will not receive treatment. They will be contacted by phone once a week to complete assessments of mood and sleep. After 4 weeks, they will cross over to the experimental BBTI group.

INTERVENTIONS:
Behavioral: Brief Behavioral Treatment for Insomnia
  Other Names: BBTI
  Arms: BBTI

SUMMARY:
The purpose of this pilot study is to obtain information about older Veterans' preferences for treatment of depression and insomnia and to pilot test the feasibility and clinical effect of Brief Behavioral Treatment for Insomnia (BBTI) BBTI for older Veterans living with Treatment Resistant Depression (TRD) and insomnia.

DETAILED DESCRIPTION:
Quantitative and qualitative methods will be used to obtain information to aid in developing treatment approaches appropriate for older Veterans with TRD and insomnia. Qualitative data will be gathered to better understand Veterans' preferences for treatment approaches, particularly relating to preference for pharmacotherapy versus augmentation with a behavioral intervention such as BBTI. Using a Randomized Controlled Trial (RCT) design, we will test whether augmentation with BBTI will be acceptable to older Veterans and improve treatment response in those whose depression has not improved with antidepressant pharmacotherapy alone and assess for an association between preference and treatment response. Our aims and hypotheses are:

Aim 1: To characterize the depression, insomnia, and relevant clinical and neuropsychiatric characteristics of older Veterans with TRD.

H1a: In Veterans with TRD, Antidepressant History Form (ATHF) scores will have a positive association with Montgomery-Asberg Depression Rating scale (MADRS) scores.

H1b: In Veterans with TRD, MADRS scores will have a positive association with Insomnia Severity Index (ISI) scores.

Aim 2: Perform qualitative interviews in older Veterans to collect information about their views of their depression and insomnia and attitudes and preferences for treatment of both depression and insomnia.

Aim 3: To examine the feasibility of using BBTI to treat Veterans with TRD and insomnia.

H3a: Use of BBTI will be feasible in older adults with TRD as defined by acceptability and retention.

Aim 4: To determine if antidepressant augmentation with BBTI leads to improvement in scores on MADRS and ISI scales in older Veterans receiving BBTI versus those receiving only antidepressant optimization.

H4a: Augmentation with BBTI will improve both PHQ-9 and ISI scores relative treatment with antidepressant alone.

ELIGIBILITY:
* Inclusion Criteria:

  * Age ≥ 60
  * Diagnosis of Major Depressive Disorder (MDD)
  * Diagnosis of Insomnia Disorder
  * Must have failed ≥ 1 antidepressant trial
* Exclusion Criteria:

  * Lifetime/current Bipolar I/II diagnosis
  * Lifetime/current Schizophrenia Spectrum Disorder diagnosis
  * Substance Use Disorder within past 3 months
  * High Suicide Risk that cannot be safely managed
  * Untreated Obstructive Sleep Apnea (OSA)
  * Restless Legs Syndrome
  * Rapid Eye Movement (REM) Sleep Behavior Disorder
  * Active OR untreated Post Traumatic Stress Disorder (PTSD)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
PHQ-9 ( depression) | 8 weeks
ISI score ( insomnia) | 8 weeks

SECONDARY OUTCOMES:
Short Form Survey (SF-12) SF-12 ( quality of life) | 8 weeks
Emotional Closeness Questionnaire ( ECQ) | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided